CLINICAL TRIAL: NCT05015270
Title: Identification of Peripheral Blood Biomarkers for Prediction of Coronary Artery Disease Confirmed by Coronary Angiography
Brief Title: Correlation of Biomarkers With the Presence and Severity of Coronary Artery Disease
Acronym: PREDICTION-NJ
Status: Completed | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Director of Cardiology and Cath Lab, Vice President of Nanjing First Hospital, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: NMU20211033
Record Dates: First submitted 2021-08-18; First posted 2021-08-20 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease
Keywords: Biomarkers, Coronary artery disease, Disease burden, Clinical events
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Peripheral blood will be collected from all patients after informal consent is obtained
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Less disease group: Patients with coronary artery diameter stenosis <70% confirmed by coronary angiography;
  Patients will be treated using guideline recommended medications or percutaneous coronary intervention at physician's discretion
  Interventions: Diagnostic Test: Medications or percutaneous coronary intervention
- Severe disease group: Patients with coronary artery stenosis ≥70% confirmed by coronary angiography;
  Patients will be treated using guideline recommended medications or percutaneous coronary intervention at physician's discretion
  Interventions: Diagnostic Test: Medications or percutaneous coronary intervention

INTERVENTIONS:
Diagnostic Test: Medications or percutaneous coronary intervention — In this study, we will for the first analyze the correlation of proteins concentration with coronary artery disease burden. Next, the prediction of proteins for one-year clinical events will be further analyzed
  Other Names: Percutaneous coronary intervention

SUMMARY:
The development of coronary artery disease is multifactorial. Peripheral blood biomarkers paly an important role in the prediction of coronary artery disease. However, the identification of those biomarkers and their correlation with the presence and severity of coronary artery disease are unclear. The present study aims to identify the differentially expressed biomarkers from peripheral blood between normal population and patients with different disease burden confirmed by coronary angiography, and to analyze the correlation of those biomarkers with the severity of coronary artery disease. Finally, the prediction of biomarkers for clinical events.

DETAILED DESCRIPTION:
This study includes three parts:

1. Part 1 (Pilot analysis): 30 normal people and 30 patients with at least one epicardial coronary artery disease confirmed by angiography will be included. 10 ml peripheral blood from arterial sheath (just before angiography) will be collected in each subject. Proteomics analyses are performed in order to obtain the differentially expressed proteins (coded by Proteins 1-x.
2. Part 2 (Training group): Differentially expressed Proteins 1-x are measured and compared between patients with diameter stenosis <70% (n=100) vs. with diameter stenosis ≥ 70%(n=100), respectively. Finally, Proteins 1-y from Proteins 1-x will be identified. Subgroups stratified by single-, double-, and triple-vessel disease will be performed.
3. Part 3 (Validation group): The difference in blood concentration of Proteins 1-y between patients with different disease burden will be further analyzed: patients with diameter stenosis <70% (n=200) vs. diameter stenosis ≥70% (n=200), respectively. Subgroups stratified by single-, double-, and triple-vessel disease will be performed.

ELIGIBILITY:
Inclusion Criteria:

* For Pilot study, both health and patients with at least one epicardial coronary artery disease are included
* For both Training group and Validation group, patients must have at least one epicardial coronary artery disease
* Left ventricular ejection fraction > 30%
* Stable or unstable angina
* Myocardial infarction older than 1 month
* No active inflammation
* No scheduled non-cardiac surgery within 12 months
* eGFR > 30 ml/min/m2
* Patients agree to participate in this study

Exclusion Criteria:

* Severe liver dysfunction
* Blood platelet count <100 x 109/L
* Cancer
* On dialysis
* Pulmonary hypertension (defined as mean pulmonary arterial pressure > 25 mmHg and pulmonary vessel resistance > 3.0 Woods Unit)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In geneal, the traditional risk factors for coronary artery disease (including age, sex, hypertension, diabetes, dyslipidemia, peripheral artery disease, smoker, fat, etc.) will be comparble between three groups (case-control).
Sampling Method: Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Correlation of biomarkers with coronary artery disease burden | 12 months
  We will analyze the differential level of proteins in peripheral blood between three groups. As a result, the correlation between biomarkers with disease burden will analyzed.

SECONDARY OUTCOMES:
Clinical events | 12 months
  Clinical events are a composite of cardiac death, myocardial infarction, revascularization, and stroke at one-year since coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang M Chen, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
No share IPD with others